CLINICAL TRIAL: NCT05857111
Title: Observational Prospective Study, to Validate the Effectiveness of CELBREA® Compared to the Detection Results in Symptomatic Women or Those With Diagnostic Doubt (DETECT-BH)
Brief Title: Effectiveness Validation of CELBREA® in Symptomatic Women or With Diagnostic Doubt of Breast Pathology (DETECT-BH)
Acronym: DETECT-BH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Jose Ignacio Sánchez (Other)
Collaborators: Welwaze Medical Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Jose Ignacio Sánchez, Head of Breast Unit - Hospital Universitario La Paz - Madrid - Spain, Instituto de Investigación Hospital Universitario La Paz
Organization: Instituto de Investigación Hospital Universitario La Paz (Other)
Other Study IDs: PI-5330; 2022.296 (Other: Hospital Universitario La Paz)
Record Dates: First submitted 2023-04-25; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Breast Disease; Benign Breast Disease; Breast Cancer
Keywords: breast symptoms; diagnostic doubt; Celbrea; Breast Thermal Activity Indicator
MeSH Terms: conditions — Breast Diseases; Cystic Fibrosis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study population: An estimate of 255 adult women (≥ 18 years old) who come to consult at the Breast Pathology Unit of La Paz Hospital (Madrid, Spain), because of discomfort, breast symptoms, or because they have been sent for specialized evaluation because of a diagnostic doubt will be included.
  Interventions: Device: Celbrea

INTERVENTIONS:
Device: Celbrea — The test with the CELBREA® device will be added to the routine screening according to the protocols of the health facility.
  Other Names: Breast Thermal Activity Indicator

SUMMARY:
This is an observational, prospective, and transversal study, designed to evaluate the effectiveness of CELBREA® in women from the local community coming to consult at the Breast Pathology Unit of La Paz Hospital (Madrid, Spain), because of discomfort, breast symptoms, or because they have been sent for specialized evaluation because of a diagnostic doubt, providing actualized data on the effectiveness of the device within the context of the real-world scenario. Because of its transverse nature, the observation period will be limited to the necessary amount of time to perform the initial consult, additional tests when prescribed by the physician, and the CELBREA® test.

ELIGIBILITY:
INCLUSION CRITERIA

1. Women ≥ 18 years old coming to consult at the Breast Pathology Unit of La Paz Hospital (Madrid, Spain), because of:

   * Discomfort or breast symptoms including, but not limited to, signs or symptoms detected through a self-examination, changes of color or shape in the nipple, nipple discharge, change of appearance or color of breast skin, lumps, etc.
   * Refered for evaluation because of diagnostic doubt.
2. Capable of following the instructions necessary for the study.
3. Have signed the informed consent form.

EXCLUSION CRITERIA:

1. Women who are pregnant or lactating at the time of the study.
2. Women suffering from one of the following breast pathologies:

   * Personal history of breast cancer, previous or current.
   * Current chemotherapy or radiotherapy for any type of cancer.
   * History of breast surgery (reductive, reconstructive, mastectomy, lumpectomy, and others).
   * Fever.
   * Swelling or local infections on the breasts.
   * Open wounds in breast skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An estimate of 255 adult women (≥ 18 years old) who come to consult at the Breast Pathology Unit of La Paz Hospital (Madrid, Spain), because of discomfort, breast symptoms, or because they have been sent for specialized evaluation because of a diagnostic doubt will be included.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-07-07 (Estimated)

PRIMARY OUTCOMES:
Effectiveness defined as sensitivity, specificity, positive and negative predictive values, positive and negative probability quotients, and accuracy using Detection Results as comparator. | Through study completion, an average of 1 year
  Detection Result (DR): it is defined as the absence or presence of a breast pathology (benign or malignant).
  Positive DR: a DR will be labeled as positive (Positive DR) when the presence (diagnosis) of a breast pathology has been verified (benign or malignant).
  Negative DR: a DR will be labeled as negative (Negative DR) when the absence of breast pathologies has been verified.
  Significant Reading (CELBREA® test): A difference of 4 columns or more between corresponding segments is considered significant.
  Non-significant reading (CELBREA® test): a difference of 3 columns or less in any section between corresponding segments is considered non-significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain